CLINICAL TRIAL: NCT02586441
Title: Evaluation of EEG With Respect to the Change of Depth of Anesthesia
Brief Title: Evaluation of EEG With Respect to the Change of Depth of Anesthesia During General Anesthesia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Joonchul Jang, Resident, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MD11004
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Last update posted 2015-11-04 (Estimated); Status verified 2015-11

CONDITIONS: Anesthesia
Keywords: Bispectral index (BIS); EEG; Depth of anesthesia
MeSH Terms: interventions — Electroencephalography; Propofol; Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Electroencephalography (Experimental): 1. Standard monitoring included electrocardiogram, noninvasive arterial blood pressure, pulse oximetry, and BIS-VISTATM sensor at OR.
  2. Raw EEG in a steady state was collected for 5 minutes.
  3. Anesthesia was induced with intravenous 1% propofol (1.5-2.5 mg/kg) and rocuronium bromide (0.6 mg/kg)
  4. Mechanical ventilation was initiated
  5. Anesthesia was maintained with desflurane at an end-tidal concentration of 6-7 %, with a fraction of inspired oxygen of 0.5 (fresh gas flow; O2 1.5 L/min and air 2.5 L/min).
  6. On completion of the surgery, all anesthetic gases were discontinued and the FiO2 was increased to 1.0.
  7. After extubation, BIS-VISTA TM monitoring was stopped.
  Interventions: Device: Electroencephalography; Drug: Propofol; Drug: Rocuronium bromide

INTERVENTIONS:
Device: Electroencephalography — Raw EEG signals were acquired at a sampling rate of 128Hz using a BIS-VISTATM monitor and was measured during all anesthetic period.
Drug: Propofol — intravenous 1% propofol (1.5-2.5 mg/kg)
  Other Names: Fresofol MCT 1%
Drug: Rocuronium bromide — intravenous rocuronium bromide (0.6 mg/kg)
  Other Names: Esmerone

SUMMARY:
The BIS Index, one of the VISTA Monitor output parameters, may be used as an aid in monitoring the effects of certain anesthetic agents;and its usage with certain anesthetic agents may be associated with a reduction in primary anesthetic use and a reduction in emergence and recovery time.

However, this equipment does not give the proper anesthetic depth index is a number of experimental results have been reported.

Therefore, the investigators study that the BIS VISTA receives an electroencephalogram (EEG) obtained through the depth of anesthesia monitors brain waves to collect statistical data, through mathematical analysis to analyze the exact correlation between the patient's brain waves and the depth of anesthesia.

DETAILED DESCRIPTION:
General anesthesia is accompanied during surgery gives a lot of satisfaction and impact on surgical outcomes of patients depending on the dose of the anesthetic, as well as operation time and intensity.

The BIS Index, one of the VISTA Monitor output parameters, may be used as an aid in monitoring the effects of certain anesthetic agents;and its usage with certain anesthetic agents may be associated with a reduction in primary anesthetic use and a reduction in emergence and recovery time.

However, this equipment does not give the proper anesthetic depth index is a number of experimental results have been reported.

Therefore, the investigators study that the BIS VISTA receives an electroencephalogram (EEG) obtained through the depth of anesthesia monitors brain waves to collect statistical data, through mathematical analysis to analyze the exact correlation between the patient's brain waves and the depth of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist[ASA] class 1-2
* written informed consent

Exclusion Criteria:

* allergy of neuromuscular blocking drugs or other medications used during general anesthesia
* known or suspected upper respiratory infection
* suspected difficult tracheal intubation
* Uncontrolled Hypertension
* known or suspected psychologic disorder
* known or suspected significant renal dysfunction
* known or suspected severe hepatic dysfunction
* known or suspected significant cardiovascular dysfunction

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
EEG acquisition | From 5minutes before induction to extubation
  Raw EEG signals were acquired at a sampling rate of 128Hz using a BIS-VISTATM monitor and was measured during intraoperative period.
  Transferring the raw EEG signal obtained from BIS VISTA monitor to a computer, the data is processed using MATLAB

CONTACTS AND LOCATIONS:
Overall Officials: Hyub Huh, M.D, Principal Investigator — Anesthesia and Pain medicine department, Korea University Anam Hospital

REFERENCES:
- [Result] Yoon YG, Kim TH, Jeong DW, Park SH. Monitoring the depth of anesthesia from rat EEG using modified Shannon entropy analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:4386-9. doi: 10.1109/IEMBS.2011.6091088. PMID 22255311